CLINICAL TRIAL: NCT04201587
Title: The Preliminary Effects of Henna on Chemotherapy-Induced Peripheral Neuropathy in Women Receiving Oxaliplatin Based Treatment: A Parallel Group Randomized Controlled Pilot Trial
Brief Title: The Preliminary Effects of Henna on CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Pinar Zorba Bahceli, PhD RN, Asistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/78
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy-induced peripheral neuropathy; Henna; Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henna application group (Experimental)
  Interventions: Other: Henna application
- Control group (No Intervention)

INTERVENTIONS:
Other: Henna application — Henna application was performed to the patients in the intervention group. The patient was instructed to apply henna before going to bed at night, and after waking up in the morning (for an average of 8-10 hours) was instructed to wash with only water. The patient was asked to do this application at home after the second and third chemotherapy cycles. Thus, the patient applied henna twice in total (fifteen days apart).
  Arms: Henna application group

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most common long-term toxicities of chemotherapy. Though, CIPN is one of the common symptoms encountered by oncology nurses in care of patients. For this reason, there is a need for an intervention that could decrease or prevent of CIPN.

DETAILED DESCRIPTION:
Chemotherapy-induced peripheral neuropathy (CIPN) is frequently seen in patients receiving oxaliplatin-based therapy.This parallel group randomized controlled pilot clinical trial aimed at investigating the feasibility and preliminary effect of henna on CIPN in women receiving oxaliplatin-based therapy. This trial was conducted in the chemotherapy outpatient clinic of University Hospital located in Turkey. All patients were women who received oxaliplatin-based therapy in the oncology clinic every fifteen days.

In order to calculate the sample size, it was decided to recruit 30 female patients to each group (intervention and control) using the G.Power-3.1.9.2 program. A total of 60 female patients were included in the study.

The study consists of two groups. In the intervention group, after the 2nd and 3rd chemotherapy cycles, henna application was applied to the hand-foot and toes. The control group underwent only the routine treatment.

To collect data, a personal information form and Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) were used.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older women
* Must the level of neurotoxicity is Stage II and Stage III
* Must taken at least one chemotherapy cycle and is planned to continue 2 chemotherapy cycles
* Be taking Folfox-6 chemotherapy protocol

Exclusion Criteria:

* Having an open wound and edema in the hands and feet
* Having a peripheral neuropathy due to diabetes and autoimmune diseases
* Using any complementary and alternative (CAM) treatment method to prevent peripheral neuropathy during administration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool-CIPNAT | It was filled before the 2nd, 3rd and 4th chemotherapy cycles (each cycle is 15 days). Change from baseline Chemotherapy-Induced Peripheral Neuropathy Assessment Tool scores at 6 weeks.
  It was developed by Tofthagen et al. (2011) to evaluate chemotherapy-induced peripheral neuropathy. It consists of two sections. The first section concerns nine symptoms; the severity of these symptoms, the possibility of an emotional problem occurring, and the incidence rate of these symptoms are evaluated. The first six questions in this section constitute the sensory symptoms, and the seventh, eighth and ninth questions constitute the subdimensions of motor symptoms. In the second section, fourteen (sensory and motor) activities were evaluated, including whether they were affected by the symptoms. The total score to be obtained from the scale is between 0 and 279. High scores indicate severe symptoms, high rate of incidence, many emotional problems and limitations on daily life activities.It was tested for validity and reliability on Turkish population by Kutluturkan et al. (2017), with Cronbach's alpha reliability coefficient of 0.95.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Arslan, PhD, Principal Investigator — Department of Internal Medicine Nursing, Faculty of Nursing, Selcuk University,Konya/Turkey
Locations (1):
- Selcuk University Faculty of Nursing, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No